CLINICAL TRIAL: NCT04429776
Title: Tapering of Biologics in Inflammatory Arthritis Patients in Remission
Acronym: TAPER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Anne Barton, Clinical Professor of Rheumatology, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 281569
Record Dates: First submitted 2020-06-05; First posted 2020-06-12 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic

STUDY DESIGN:
Intervention Model Description: 50 Participants: randomised 1:1 to either feedback of test results to treating clinician or no feedback to treating clinician (25 participants each arm)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feedback Arm (Experimental): Trough blood samples taken and analysed at baseline, 6m and 12m. Results fed back to recruiting clinical team who can choose to use these to influence their tapering decisions.
  Interventions: Diagnostic Test: Drug level testing with feedback provided
- No Feedback Arm (Active Comparator): Trough blood samples taken and analysed at baseline, 6m and 12m. Results not fed back to recruiting clinical team.
  Interventions: Diagnostic Test: Drug level testing with no feedback provided

INTERVENTIONS:
Diagnostic Test: Drug level testing with feedback provided — Feedback about drug levels in blood provided to participant's site
  Other Names: Anti-drug antibody testing
  Arms: Feedback Arm
Diagnostic Test: Drug level testing with no feedback provided — Testing drug levels in blood but feedback not provided to participant's site
  Other Names: Anti-drug antibody testing
  Arms: No Feedback Arm

SUMMARY:
Rheumatoid arthritis (RA) and Psoriatic Arthritis (PsA) are types of inflammatory arthritis. They are disabling conditions caused by inflammation in joints that can lead to pain, stiffness, fatigue and joint damage. There is currently no cure but treatment is aimed at reducing joint inflammation. Some of the most promising new therapies work by interfering with the binding of a molecule called tumour necrosis factor (TNF). In recent years, new anti-TNF drugs (such as adalimumab, etanercept and certolizumab) have been developed that block the action of TNF and reduce this inflammation. These drugs are very effective in controlling inflammation for many patients whose arthritis has not responded to other therapies. Some patients can take these medications for a long time. If a patient is stable on their rheumatoid arthritis biologic or biosimilar, tapering the drug is often considered.

The investigators are planning to look at drug level and anti-drug antibody testing to guide anti-TNF tapering (reducing) decisions in UK patients with RA who have stable, reduced arthritis symptoms. The investigators think that measuring these drug levels and anti-drug antibodies in blood samples will be useful for guiding this process, but the investigators can't be sure. It is important to do this safely so the patient doesn't experience a flare of their disease symptoms. The study will be used to determine whether a much larger study to assess the usefulness of these measurements would be achievable.

This study will assess whether measuring biomarkers (measurable substances in the blood) that may affect a patient's response to treatment.

If a patient are eligible to take part, they will be randomly allocated to one of the following groups;

* Their Doctor receiving information and treatment advice based on their blood results or
* Their Doctor not receiving this information

DETAILED DESCRIPTION:
Participants will be randomly allocated to feedback of their drug levels / antidrug antibody status to their consultant prior to tapering, or not, in a 1:1 ratio.

* Those participants randomised to the group where no feedback is required will have their dosing interval doubled (from 2 to 4 weeks for certolizumab and adalimumab; from 1 to 2 weeks for etanercept).
* For participants randomised to the arm where results are received by the treating clinician, advice will accompany the results. It will be made clear that this is advice only and that the ultimate treatment decisions rest with the treating clinician.

Patients would be recruited at the point at which the decision is made to begin tapering their biologic.

The NHS site teams will be informed which arm of the study the participant has been randomised to, as they will be made aware of patient test results. Participants will not be blinded to which intervention they receive. University of Manchester Researchers undertaking the laboratory tests and those entering study data will be blinded.

The consent form, registration form, baseline CRF and baseline participant questionnaire should then be returned to the study coordinator at CfMR in the pre-paid packaging provided.

A baseline DAS28 score must be provided. This should be from no more than a month before the date of consent. If this cannot be provided the patient is not eligible to take part.

Recruiting teams can start to taper the patient's medication immediately after consent on to the TAPER trial.

Blood samples will be taken at the following time points;

* Baseline (at the point of consent, when the decision to taper is made)
* 6 months after tapering starts
* 12 months after tapering starts Participants in TAPER will need to have their blood samples taken the day before their next anti-TNF injection date. This means the participant will have to come in to their hospital sites at these time points for their sample. Sites will be provided with blood kits for this. These will include a phlebotomy letter, just in case the participant needs to go to a different hospital department to have their bloods taken. These will be returned to the University of Manchester is the pre-paid postage boxes provided.

The researchers would like each of the follow-up visits to occur as closely to the 6 month and 12 month time points as possible. However, the researchers will accept the following visit windows;

• 6 and 12 month time points; +/- 1 month The University of Manchester will return the blood results to site for participants randomised to the arm where results are returned. This will be sent via email with appropriate treatment advice, as per the information in section 4 within 4 weeks of sample receipt. The site team will receive these results by letter in advance of the follow-up visit and will have the opportunity to discuss these with the Chief Investigator, Prof. Anne Barton, in advance of the visit if required. For participants in the control arm (no feedback of results), the blood samples will be collected and tested in the same way but results will not be provided to the treating clinician.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have RA according to the American College of Rheumatology (ACR) 1987 or 2010 criteria
2. Patients must be willing and able to participate in the study (including follow up visits and providing blood samples) after providing informed consent.
3. Patients must currently be on stable treatment a one of the following single anti-TNF agents Adalimumab, Etanercept or Certolizumab. They must have been taking this biologic/ biosimilar therapy for a minimum of 12 months
4. Patients must be in remission with a DAS28 CRP of less than or equal to 2.6.
5. A DAS28 score must be provided at baseline. This must have been taken within the month before study recruitment. If this DAS score is not available, the patient is not eligible to take part.
6. Consultant must be looking to taper patient's standard care medication
7. Aged 18 years or over

Exclusion Criteria:

1. Anyone who has switched anti-TNF agent in the last 12 months
2. Anyone without a recent DAS score (within the previous month)
3. Anyone taking any anti-TNF therapy that isn't Adalimumab, Etanercept or Certolizumab.
4. Anyone who has received steroids within past 3 months (enteral, parenteral or intra-articular)
5. Anyone who is currently pregnancy, or pregnancy planned within next 6 months
6. Anyone with any planned major surgery
7. Anyone with the inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to flare | 3 years
  Time to flare

SECONDARY OUTCOMES:
Successful recruitment | 3 years
  Successful recruitment
Was biologic advice, provided in the protocol, adopted by clinicians and participants? | 3 years
  Adoption of biologic advice by clinicians and participants; assessed by end of study questionnaires
Participant withdrawal rate | 3 years
  Participant withdrawal rate
Participant acceptability, via the feedback form | 3 years
  Participant acceptability, via the feedback form
Participant reported outcome measures recorded in the participant questionnaire booklet. | 3 years
  Participant reported outcome measures recorded in the participant questionnaire booklet.

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University Hospitals NHS Foundation Trust, Manchester, North West, United Kingdom

IPD SHARING:
Plan to Share IPD: No